CLINICAL TRIAL: NCT01963962
Title: A Prospective Trial of the Copper T380 IUD or Oral Levonorgestrel and the Levonorgestrel IUD Initiated With Emergency Contraception
Brief Title: Study of the Copper IUD or Oral Levonorgestrel and the Levonorgestrel IUD for Women Seeking Emergency Contraception
Acronym: COLIEC
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, M.D., University of Utah
Other Study IDs: 50483
Record Dates: First submitted 2013-10-11; First posted 2013-10-17 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Emergency Contraception
Keywords: Emergency contraception; Levonorgestrel IUD; Copper IUD; Oral Levonorgestrel
MeSH Terms: interventions — Intrauterine Devices, Copper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine to test for progesterone and/or pregnandiol
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Copper IUD: Women selecting the copper IUD for emergency contraception and to use for contraception after
  Interventions: Drug: Copper IUD
- Levonorgestrel IUD: Women who select oral levonorgestrel for emergency contraception and begin the levonorgestrel IUD for ongoing contraception at the same time.
  Interventions: Drug: Levonorgestrel IUD

INTERVENTIONS:
Drug: Copper IUD
  Other Names: Paragard IUD
  Groups: Copper IUD
Drug: Levonorgestrel IUD
  Other Names: Mirena IUD
  Groups: Levonorgestrel IUD

SUMMARY:
The purpose of this study is to see how often women who come to a family planning clinic for emergency contraception, the morning after pill, are willing to use either the copper IUD or the levonorgestrel IUD. The investigators will also see if pregnancies occur in those choosing the levonorgestrel IUD and if people continue to use the IUD for 1 year.

DETAILED DESCRIPTION:
Widely available oral levonorgestrel (LNG) for emergency contraception (EC) has not reduced unplanned pregnancy rates. However, our study of the copper T380 IUD vs. oral LNG for EC showed lower pregnancy rates 12 months after presenting for EC in the copper IUD group. Because there is a strong preference for the LNG IUD among women offered the IUD, the objective of this research project is to initiate investigation into, and use of the LNG IUD in the setting of EC. Our experienced team of EC researchers proposes the following aims to provide needed information in this understudied area:

Aim 1: To assess uptake of the LNG IUD vs. the copper IUD among women presenting for EC exposed to standardized counseling.

Aim 2: Gather baseline data on one-year continuation and pregnancy rates from women initiating the LNG IUD vs. the copper T380 IUD when presenting for EC.

Aim 3: Assess willingness of women presenting for EC to participate in a future randomized controlled trial comparing the LNG IUD vs. the copper T380 IUD for EC.

The study aims will be accomplished with a prospective observational trial of women who choose either method of EC. The investigative team will recruit 180 women who present for EC at two participating family planning clinics and follow study participants for 12 months. This project will compare continuation and pregnancy rates between LNG and copper IUD users in the year following presentation for EC. This proposal is another aspect in our growing research program offering highly effective contraception at the time of EC presentation. Results of this project will direct future study in this area aimed at reducing population unplanned pregnancy rates among EC users with the potential to inform a future RCT of the LNG vs. copper IUD for EC.

ELIGIBILITY:
Inclusion Criteria:1. Between 18-35 years old

2. In need of EC (had unprotected intercourse within 120 hours - 5 days)

3. Desire to prevent pregnancy for 1 year

4. Fluent in English and/or Spanish

5. Have a regular menstrual cycle (24-35 days)

6. Know their last menstrual period (+/-3 days)

7. Be willing to comply with the study requirements

8. Participants current preferred phone number must be functioning at the time of study entry and will be tested prior to enrollment

-

Exclusion Criteria:

* 1. Current pregnancy

  2. Breastfeeding

  3. Intrauterine infection within the past 3 months

  4. Sterilization

  5. Already have an IUD or contraceptive implant (Implanon) in place

  6. Vaginal bleeding of unknown etiology

  7. Known Gonorrhea or Chlamydia infection in the last 30 days (unless successfully treated at least 7 days prior to study entry)

  8. Allergy to LNG (for LNG IUD patients)

  9. Allergy to copper or Wilson's disease (for Copper IUD patients)

  10. Known abnormalities of the uterus that distort the uterine cavity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women presenting for emergency contraception to family planning clinics in Salt Lake City, UT
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates in first month after IUD insertion | 4 weeks
  Participants will have a urine pregnancy test at the clinic. They will also be given a home urine pregnancy test to check if they are not able to return to clinic and will give results by phone or electronic communication.

SECONDARY OUTCOMES:
1 Year IUD continuation rates | 1 year
  IUD continuation rates will be compared between those who selected the copper IUD and thos who selected the levonorgestrel IUD

OTHER OUTCOMES:
Willingness to be randomized to either the copper or levonorgestrel IUD for emergency contraception. | At enrollment
  We will query all participants to see if they would be willing to participate in a randomized study where the type of IUD (copper vs. levonorgestrel) was chosen at random.

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator — University of Utah
Locations (1):
- Planned Parenthood Association of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Boraas CM, Sanders JN, Schwarz EB, Thompson I, Turok DK. Risk of Pregnancy With Levonorgestrel-Releasing Intrauterine System Placement 6-14 Days After Unprotected Sexual Intercourse. Obstet Gynecol. 2021 Apr 1;137(4):623-625. doi: 10.1097/AOG.0000000000004118. PMID 33706343
- [Derived] Turok DK, Sanders JN, Thompson IS, Royer PA, Eggebroten J, Gawron LM. Preference for and efficacy of oral levonorgestrel for emergency contraception with concomitant placement of a levonorgestrel IUD: a prospective cohort study. Contraception. 2016 Jun;93(6):526-32. doi: 10.1016/j.contraception.2016.01.009. Epub 2016 Mar 2. PMID 26944863